CLINICAL TRIAL: NCT04141189
Title: Comparison of Follow-up Protocols in Terms of Fetal, Neonatal and Maternal Results in Intrauterine Growth Retardation: a Randomised Controlled Trial
Brief Title: Comparison of Follow-up Protocols in Terms of Fetal, Neonatal and Maternal Results in Intrauterine Growth Retardation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BezmialemVU fetal surveillance
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Fetal Surveillance; Intrauterine Growth Restriction
Keywords: Intrauterine Growth Restriction; fetal surveillance; fetal doppler; fetal growth
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weekly (Experimental): weekly fetal surveillance
  Interventions: Procedure: weekly
- bi-weekly (twice-weekly) (Active Comparator): bi-weekly fetal surveillance
  Interventions: Procedure: bi-weekly

INTERVENTIONS:
Procedure: weekly — fetal surveillance frequency
  Arms: weekly
Procedure: bi-weekly — fetal surveillance frequency
  Arms: bi-weekly (twice-weekly)

SUMMARY:
This study will be undertaken to determine whether the frequency of fetal surveillance can be safely reduced from bi-weekly to weekly in the case of fetusus with intrauterine growth restriction.

DETAILED DESCRIPTION:
In this prospective randomized study, the cases whose fetal weight predicted by ultrasonography (USG) between the 28th and 37th weeks of gestation are below 10percentile according to the World Health Organization (WHO) normograms. The cases will be divided into two groups as group 1:weekly and group 2:bi-weekly (twice-weekly) The cases will be evaluated by fetal Doppler, amniotic fluid volume, nonstress test (NST) and maternal preeclampsia tests.Maternal severe hypertension/preeclampsia, category 3 NST, oligohydramnios (after 37 weeks amniotic fluid index <5; after 34 weeks single deepest pocket <2 cm) ,pathological doppler (before 34 weeks reverse flow in an umbilical artery , after 34 weeks absent end-diastolic flow in an umbilical artery) in cases of birth decision will be taken. Cases without the above mentioned complications will be delivered between 38 weeks 3 days and 39 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 28-37 weeks pregnant women with estimated fetal weight below 10 percentile
* singlton pregnancy

Exclusion Criteria:

* maternal preeclampsia
* maternal systemic disease (pregestational diabetes, gestational diabetes mellitus a2, antiphospholipid antibody syndrome, chronic kidney disease)
* oligohydramnios (after 34 weeks amniotic fluid index <5; before 34 weeks single deepest pocket <2 cm)
* pathological doppler (high umbilical artery resistance index, absence of end-diastolic flow velocity in the umbilical artery, reverse flow in the umbilical artery, brain sparing effect in middle cerebral artery, abnormal ductus venosus flow)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 206 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
neonatal hospital stay | 3 months
  duration of neonatal hospital stay (days)

SECONDARY OUTCOMES:
antenatal hospital stay | 3 months
  duration of antenatal hospital stay (days)

OTHER OUTCOMES:
gestational age at delivery | 24 hours
  gestational age at delivery as days (e.g. 261days)
neonatal hospital stay | 3 months
  duration of neonatal hospital stay (days)
acidosis | 24 hours
  fetal acidosis (normal cord-blood pH ranges from 7.14 to 7.4 during labor, values below 7.14 are considered to be acidosis)
perinatal death | 3 months
  The number of perinatal deaths. Perinatal death is a fetal death (stillbirth) or an early neonatal death (first 24 hours after birth)
cesarean delivery | 24 hours
  The number of births by cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided